CLINICAL TRIAL: NCT00318149
Title: Demonstrate the Non-inferiority in Term of Cellular Mediated Immune Response of GSK Biologicals' Influenza Candidate Vaccines Containing Various Adjuvants Administered in Elderly Population (Aged 65 Years &Amp; Older) vs Fluarix™ (Known as Alpha-Rix™ in Belgium) Administered in Adults (18-40 Years)
Brief Title: Safety Study of Four Candidate Influenza Vaccines to Prevent Influenza Disease in the Elderly Population
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 104886
Record Dates: First submitted 2006-04-25; First posted 2006-04-26 (Estimated); Results first posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-02

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — fluarix

ARMS (6):
- Fluarix 18-40 Y Group (Experimental): Subjects (aged 18-40 years [Y]) received 1 dose of the Fluarix vaccine, administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Fluarix
- Fluarix ≥65 Y Group (Experimental): Subjects (aged ≥ 65 years) received 1 dose of the Fluarix vaccine, administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Fluarix
- Fluarix-AS25 Group (Experimental): Subjects (aged ≥ 65 years) received 1 dose of the Fluarix vaccine adjuvanted with AS25, administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Fluarix-AS25
- Fluarix-AS50 Group (Experimental): Subjects (aged ≥ 65 years) received 1 dose of the Fluarix vaccine adjuvanted with AS50, administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Fluarix-AS50
- Fluarix- AS01B Group (Experimental): Subjects (aged ≥ 65 years) received 1 dose of the Fluarix vaccine adjuvanted with AS01B, administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Fluarix-AS01B
- Fluarix- AS01E Group (Experimental): Subjects (aged ≥ 65 years) received 1 dose of the Fluarix vaccine adjuvanted with AS01E, administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Fluarix-AS01E

INTERVENTIONS:
Biological: Fluarix — 1 dose administered intramuscularly in the deltoid region of the non-dominant arm
  Other Names: GlaxoSmithKline Biologicals' licensed influenza vaccine
  Arms: Fluarix 18-40 Y Group; Fluarix ≥65 Y Group
Biological: Fluarix-AS25 — 1 dose administered intramuscularly into the deltoid region of the non-dominant arm
  Other Names: Fluarix vaccine adjuvanted with AS25
  Arms: Fluarix-AS25 Group
Biological: Fluarix-AS50 — 1 dose administered intramuscularly into the deltoid region of the non-dominant arm
  Other Names: Fluarix vaccine adjuvanted with AS25
  Arms: Fluarix-AS50 Group
Biological: Fluarix-AS01B — 1 dose administered intramuscularly into the deltoid region of the non-dominant arm
  Other Names: Fluarix vaccine adjuvanted with AS01B
  Arms: Fluarix- AS01B Group
Biological: Fluarix-AS01E — 1 dose administered intramuscularly into the deltoid region of the non-dominant arm
  Other Names: Fluarix vaccine adjuvanted with AS01E
  Arms: Fluarix- AS01E Group

SUMMARY:
As influenza vaccine efficacy is reported to be lower in elderly subjects compared to healthy adults, probably as a result of immunosenescence, there is a desire to devise ways to increase the current vaccines efficacy for this target population. Adjuvants are known to boost immune responses, thus representing one way to increase the efficacy of the current GlaxoSmithKline Fluarix™ influenza vaccine in elderly subjects. The purpose of this study is to evaluate the immunogenicity and the reactogenicity of a vaccination with four different adjuvanted GlaxoSmithKline influenza vaccines administered to elderly subjects. For immunogenicity and safety evaluations, healthy adults aged 18 to 40 years old and elderly aged 65 years and older will receive Fluarix™ and form the control groups of this trial.

ELIGIBILITY:
Inclusion Criteria:

* A male or female aged between 18 and 40 years or aged 65 years or older at the time of the vaccination.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the administration of the study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the administration of the study vaccine.
* History of confirmed influenza infection since a year from the date of previous vaccination.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination
* History of hypersensitivity to vaccines.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Acute clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the administration of the study vaccine or during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2005-10-10 (Actual); Primary Completion 2006-05-14 (Actual); Study Completion 2006-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 104886 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104886 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104886 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104886 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104886 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104886 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluarix 18-40 Y Group: Subjects (aged 18-40 years) received 1 dose of the Fluarix vaccine, administered intramuscularly in the deltoid region of the non-dominant arm.
Period: Overall Study
Arm/Group | Fluarix 18-40 Y Group | Fluarix ≥65 Y Group | Fluarix-AS25 Group | Fluarix-AS50 Group | Fluarix- AS01B Group | Fluarix- AS01E Group
Started | 75 | 50 | 75 | 75 | 75 | 75
Completed | 75 | 50 | 75 | 75 | 75 | 73
Not Completed | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluarix 18-40 Y Group | Fluarix ≥65 Y Group | Fluarix-AS25 Group | Fluarix-AS50 Group | Fluarix- AS01B Group | Fluarix- AS01E Group | Total
Number analyzed (Participants) | 75 | 50 | 75 | 75 | 75 | 75 | 425
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.9 (5.47) | 69.3 (3.31) | 69.2 (2.98) | 69.1 (3.51) | 69.5 (3.3) | 69.5 (4.06) | 61.66 (17.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 19 | 29 | 34 | 36 | 29 | 193
  Male | 29 | 31 | 46 | 41 | 39 | 46 | 232
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: Asian - Central/South Asian heritage | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Geographic ancestry: White - Caucasian/European heritage | 72 | 50 | 75 | 75 | 75 | 75 | 422
  Geographic ancestry: Other | 2 | 0 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Influenza-specific Cluster of Differentiation 4+ (CD4+) T-cells Expressing at Least 2 Markers
Description: The frequency was expressed as the geometric mean of influenza-specific CD4 T-cells, expressing at least 2 markers among CD40 Ligand (CD40L), Interleukin 2 (IL-2), Tumor Necrosis Factor-α (TNF-α) and Interferon-γ (IFN-γ ) upon in vitro stimulation.
Time Frame: At Day 21
Population: The analysis was performed on the According-To-Protocol cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity measures were available (subjects for whom assay results were available for antibodies against at least 1 study vaccine antigen component after vaccination).
Measure: Geometric Mean (Standard Deviation); unit: T-cells/million cells
Arm/Group | Fluarix 18-40 Y Group | Fluarix ≥65 Y Group | Fluarix-AS25 Group | Fluarix-AS50 Group | Fluarix- AS01B Group | Fluarix- AS01E Group
Number analyzed (Participants) | 75 | 49 | 70 | 73 | 74 | 74
T-cells/million cells | 3229.25 (1643.2) | 1646.05 (1557.22) | 3056.06 (2059.35) | 2589.31 (2110.15) | 2454.93 (1758.20) | 2428.78 (2693.71)
Statistical Analysis 1: Comparison: Fluarix 18-40 Y Group vs Fluarix-AS25 Group; Demonstration of non inferiority of the influenza adjuvanted vaccine Fluarix-AS25 administered to elderly subjects (aged 65 years and older) as compared to the licensed influenza vaccine Fluarix administered to adults (aged 18-40 years) in terms of frequency of influenza-specific CD4 T-cells producing at least 2 different cytokines (CD40L, IL-2, TNF-α or IFN-γ), 21 days post-vaccination; Test type: Non-Inferiority — Non inferiority criteria: The upper limit (UL) of the 2-sided 98.75% confidence interval (CI) on geometric mean ratio of influenza-specific T-cells (between Fluarix 18-40 Y Group and Fluarix-AS25 Group) was smaller than (<) 2.0; Geometric mean ratio = 0.9, 98.75% CI 2-sided [0.7 to 1.16]
Statistical Analysis 2: Comparison: Fluarix 18-40 Y Group vs Fluarix-AS50 Group; Demonstration of non inferiority of the influenza adjuvanted vaccine Fluarix-AS50 administered to elderly subjects (aged 65 years and older) as compared to the licensed influenza vaccine Fluarix administered to adults (aged 18-40 years) in terms of frequency of influenza-specific CD4 T-cells producing at least 2 different cytokines (CD40L, IL-2, TNF-α or IFN-γ), 21 days post-vaccination; Test type: Non-Inferiority — Non inferiority criteria: The upper limit (UL) of the 2-sided 98.75% confidence interval (CI) on geometric mean ratio of influenza-specific T-cells (between Fluarix 18-40 Y Group and Fluarix-AS50 Group) was smaller than (<) 2.0; Geometric mean ratio = 1.05, 98.75% CI 2-sided [0.71 to 1.56]
Statistical Analysis 3: Comparison: Fluarix 18-40 Y Group vs Fluarix- AS01B Group; Demonstration of non inferiority of the influenza adjuvanted vaccine Fluarix-AS01B administered to elderly subjects (aged 65 years and older) as compared to the licensed influenza vaccine Fluarix administered to adults (aged 18-40 years) in terms of frequency of influenza-specific CD4 T-cells producing at least 2 different cytokines (CD40L, IL-2, TNF-α or IFN-γ), 21 days post-vaccination; Test type: Non-Inferiority — Non inferiority criteria: The upper limit (UL) of the 2-sided 98.75% confidence interval (CI) on geometric mean ratio of influenza-specific T-cells (between Fluarix 18-40 Y Group and Fluarix-AS01B Group) was smaller than (<) 2.0; Geometric mean ratio = 1.04, 98.75% CI 2-sided [0.79 to 1.38]
Statistical Analysis 4: Comparison: Fluarix 18-40 Y Group vs Fluarix- AS01E Group; Demonstration of non inferiority of the influenza adjuvanted vaccine Fluarix-AS01E administered to elderly subjects (aged 65 years and older) as compared to the licensed influenza vaccine Fluarix administered to adults (aged 18-40 years) in terms of frequency of influenza-specific CD4 T-cells producing at least 2 different cytokines (CD40L, IL-2, TNF-α or IFN-γ), 21 days post-vaccination; Test type: Non-Inferiority — Non inferiority criteria: The upper limit (UL) of the 2-sided 98.75% confidence interval (CI) on geometric mean ratio of influenza-specific T-cells (between Fluarix 18-40 Y Group and Fluarix-AS01E Group) was smaller than (<) 2.0; Geometric mean ratio = 1.07, 98.75% CI 2-sided [0.79 to 1.44]

2. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 3 Strains of Influenza Disease
Description: Titers are presented as geometric mean titers (GMTs). The 3 flu strains assessed were A/New Caledonia (H1N1), A/New York (H3N2) and B/Jiangsu (B).
  Seropositivity was defined as a serum HI titer greater than or equal to (≥) 1:10.
Time Frame: At Day 0 and at Day 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Fluarix 18-40 Y Group | Fluarix ≥65 Y Group | Fluarix-AS25 Group | Fluarix-AS50 Group | Fluarix- AS01B Group | Fluarix- AS01E Group
Number analyzed (Participants) | 75 | 49 | 74 | 75 | 75 | 75
Titers
  A/New Caledonia, Day 0 | 20.7 [14.3 to 30.2] | 23.5 [16.2 to 34.1] | 23.9 [17.6 to 32.5] | 24.1 [18.1 to 32.3] | 33.9 [24.5 to 46.9] | 33.5 [24.5 to 45.9]
  A/New Caledonia, Day 21 | 728.4 [549.2 to 966.0] | 86.5 [58.7 to 127.4] | 151.9 [115.1 to 200.5] | 223.2 [170.5 to 292.3] | 151.4 [118.4 to 193.6] | 166.8 [130.1 to 213.9]
  A/New York, Day 0 | 16.5 [12.8 to 21.4] | 12.0 [9.2 to 15.6] | 13.0 [10.1 to 16.7] | 16.0 [12.1 to 21.2] | 15.5 [12.3 to 19.6] | 17.2 [12.9 to 22.9]
  A/New York, Day 21 | 151.3 [119.8 to 191.1] | 98.9 [65.1 to 150.3] | 249.7 [186.2 to 334.8] | 240.3 [176.0 to 328.0] | 202.5 [157.6 to 260.2] | 249.3 [181.7 to 342.0]
  B/Jiangsu, Day 0 | 25.2 [18.9 to 33.6] | 31.4 [21.8 to 45.2] | 27.7 [21.1 to 36.5] | 38.7 [27.7 to 54.0] | 39.2 [30.2 to 51.0] | 30.0 [23.2 to 38.8]
  B/Jiangsu, Day 21 | 349.5 [270.7 to 451.2] | 134.1 [100.2 to 179.4] | 237.1 [185.1 to 303.8] | 293.1 [234.1 to 366.8] | 205.4 [171.3 to 246.2] | 202.6 [161.2 to 254.6]

3. Secondary Outcome: Titers for Serum HI Antibodies Against 3 Strains of Influenza Disease
Description: Titers are presented as geometric mean titers (GMTs). The 3 flu strains assessed were A/New Caledonia (H1N1), A/New York (H3N2) and B/Jiangsu (B).
  Seropositivity was defined as a serum HI titer of ≥ 1:10.
Time Frame: At Day 90 and Day 180
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for persistence included all subjects from the ATP cohort for immunogenicity who had not received any medication or vaccine forbidden by the protocol during the study period and who had available assay results for at least 1 tested antigen at the Day 90 or Day 180 time points.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Fluarix 18-40 Y Group | Fluarix ≥65 Y Group | Fluarix-AS25 Group | Fluarix-AS50 Group | Fluarix- AS01B Group | Fluarix- AS01E Group
Number analyzed (Participants) | 75 | 49 | 74 | 74 | 74 | 74
Titers
  A/New Caledonia, Day 90 | 496.4 [370.1 to 665.7] | 76.7 [54.1 to 108.8] | 94.2 [74.7 to 118.8] | 135.3 [102.4 to 178.7] | 97.4 [78.1 to 121.4] | 105.9 [84.3 to 133.0]
  A/New Caledonia, Day 180: number analyzed (Participants) | 74 | 49 | 74 | 74 | 74 | 73
  A/New Caledonia, Day 180 | 354.7 [260.3 to 483.5] | 62.9 [45.4 to 87.1] | 66.9 [53.3 to 84.1] | 89.1 [67.2 to 118.2] | 70.5 [56.5 to 87.9] | 81.9 [65.1 to 103.0]
  A/New York, Day 90 | 130.5 [100.8 to 168.9] | 60.7 [41.4 to 89.1] | 99.2 [75.2 to 131.0] | 116.4 [88.6 to 153.0] | 93.3 [73.2 to 119.0] | 114.8 [85.1 to 154.8]
  A/New York, Day 180: number analyzed (Participants) | 74 | 49 | 74 | 74 | 74 | 73
  A/New York, Day 180 | 96.5 [73.5 to 126.6] | 43.8 [30.2 to 63.7] | 66.3 [50.5 to 87.1] | 71.8 [55.6 to 92.7] | 59.5 [46.8 to 75.6] | 70.4 [53.0 to 93.4]
  B/Jiangsu, Day 90 | 208.2 [161.0 to 269.3] | 131.3 [98.1 to 175.8] | 145.6 [110.7 to 191.6] | 213.0 [173.0 to 262.1] | 147.1 [120.7 to 179.2] | 144.2 [116.6 to 178.4]
  B/Jiangsu, Day 180: number analyzed (Participants) | 74 | 49 | 74 | 74 | 74 | 73
  B/Jiangsu, Day 180 | 140.3 [109.0 to 180.5] | 94.5 [69.2 to 129.0] | 91.6 [71.4 to 117.6] | 128.0 [102.6 to 159.8] | 111.0 [88.3 to 139.6] | 91.4 [74.3 to 112.3]

4. Secondary Outcome: Number of Seroconverted Subjects Against 3 Strains of Influenza Disease
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination titer <1:10 and a post-vaccination titer ≥1:40 or a pre-vaccination titer ≥1:10 and at least a four-fold increase in post-vaccination titer. The 3 flu strains assessed were A/New Caledonia (H1N1), A/New York (H3N2) and B/Jiangsu (B).
Time Frame: At Day 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 18-40 Y Group | Fluarix ≥65 Y Group | Fluarix-AS25 Group | Fluarix-AS50 Group | Fluarix- AS01B Group | Fluarix- AS01E Group
Number analyzed (Participants) | 75 | 49 | 74 | 75 | 75 | 75
Participants
  A/New Caledonia (H1N1) | 58 | 15 | 41 | 56 | 36 | 39
  A/New York (H3N2) | 57 | 34 | 67 | 62 | 64 | 60
  B/Jiangsu (B). | 61 | 22 | 54 | 50 | 49 | 53

5. Secondary Outcome: Number of Seroconverted Subjects Against 3 Strains of Influenza Disease
Description: as for outcome 4
Time Frame: At Day 90 and Day 180
Population: The analysis was performed on the According-To-Protocol cohort for persistence included all subjects from the ATP cohort for immunogenicity who had not received any medication or vaccine forbidden by the protocol during the study period and who had available assay results for at least 1 tested antigen at the Day 90 or Day 180 time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 18-40 Y Group | Fluarix ≥65 Y Group | Fluarix-AS25 Group | Fluarix-AS50 Group | Fluarix- AS01B Group | Fluarix- AS01E Group
Number analyzed (Participants) | 75 | 49 | 74 | 74 | 74 | 74
Participants
  A/New Caledonia, Day 90 | 56 | 16 | 32 | 38 | 25 | 28
  A/New Caledonia, Day 180: number analyzed (Participants) | 74 | 49 | 74 | 74 | 74 | 73
  A/New Caledonia, Day 180 | 54 | 10 | 20 | 25 | 16 | 15
  A/New York, Day 90 | 55 | 29 | 56 | 55 | 47 | 48
  A/New York, Day 180: number analyzed (Participants) | 74 | 49 | 74 | 74 | 74 | 73
  A/New York, Day 180 | 48 | 17 | 40 | 40 | 35 | 35
  B/Jiangsu, Day 90 | 53 | 16 | 38 | 44 | 33 | 44
  B/Jiangsu, Day 180: number analyzed (Participants) | 74 | 49 | 74 | 74 | 74 | 73
  B/Jiangsu, Day 180 | 45 | 16 | 28 | 33 | 26 | 25

6. Secondary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against 3 Strains of Influenza Disease
Description: The seroconversion factor (SCF) was defined as the fold change in serum Hemagglutination Inhibition (HI) geometric mean titers (GMTs) post vaccination compared to pre-vaccination time point. The 3 flu strains assessed were A/New Caledonia (H1N1), A/New York (H3N2) and B/Jiangsu (B).
Time Frame: At Day 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Fluarix 18-40 Y Group | Fluarix ≥65 Y Group | Fluarix-AS25 Group | Fluarix-AS50 Group | Fluarix- AS01B Group | Fluarix- AS01E Group
Number analyzed (Participants) | 75 | 49 | 74 | 75 | 75 | 75
Fold change
  A/New Caledonia | 35.1 [21.9 to 56.4] | 3.7 [2.4 to 5.7] | 6.4 [4.5 to 9.0] | 9.2 [6.4 to 13.3] | 4.5 [3.3 to 6.1] | 5.0 [3.6 to 6.9]
  A/New York | 9.2 [7.1 to 11.8] | 8.2 [5.7 to 11.8] | 19.2 [14.6 to 25.3] | 15.0 [11.2 to 20.2] | 13.1 [10.0 to 17.1] | 14.5 [10.4 to 20.2]
  B/Jiangsu | 13.9 [10.1 to 19.1] | 4.3 [3.0 to 6.1] | 8.5 [6.5 to 11.2] | 7.6 [5.6 to 10.2] | 5.2 [4.2 to 6.5] | 6.7 [5.1 to 8.9]

7. Secondary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against 3 Strains of Influenza Disease
Description: as for outcome 6
Time Frame: At Day 90 and Day 180
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Fluarix 18-40 Y Group | Fluarix ≥65 Y Group | Fluarix-AS25 Group | Fluarix-AS50 Group | Fluarix- AS01B Group | Fluarix- AS01E Group
Number analyzed (Participants) | 75 | 49 | 74 | 74 | 74 | 74
Fold change
  A/New Caledonia, Day 90 | 23.9 [15.6 to 36.8] | 3.3 [2.3 to 4.7] | 3.9 [3.0 to 5.2] | 5.7 [4.0 to 8.1] | 2.9 [2.2 to 3.9] | 3.1 [2.3 to 4.1]
  A/New Caledonia, Day 180: number analyzed (Participants) | 74 | 49 | 74 | 74 | 74 | 73
  A/New Caledonia, Day 180 | 17.1 [11.2 to 26.0] | 2.7 [1.9 to 3.7] | 2.8 [2.2 to 3.6] | 3.7 [2.6 to 5.4] | 2.1 [1.6 to 2.8] | 2.4 [1.8 to 3.2]
  A/New York, Day 90 | 7.9 [6.3 to 10.0] | 5.1 [3.7 to 7] | 7.6 [6.1 to 9.6] | 7.3 [5.7 to 9.2] | 6.2 [4.8 to 7.9] | 6.6 [5.0 to 8.6]
  A/New York, Day 180: number analyzed (Participants) | 74 | 49 | 74 | 74 | 74 | 73
  A/New York, Day 180 | 5.8 [4.7 to 7.3] | 3.7 [2.7 to 4.9] | 5.1 [4.2 to 6.3] | 4.5 [3.5 to 5.8] | 3.9 [3.1 to 5.0] | 4.1 [3.2 to 5.3]
  B/Jiangsu, Day 90 | 8.3 [6.2 to 11.0] | 4.2 [3 to 5.9] | 5.3 [4.2 to 6.6] | 5.6 [4.3 to 7.2] | 3.7 [3 to 4.6] | 4.8 [3.7 to 6.1]
  B/Jiangsu, Day 180: number analyzed (Participants) | 74 | 49 | 74 | 74 | 74 | 73
  B/Jiangsu, Day 180 | 5.4 [4.3 to 7.0] | 3 [2.2 to 4.1] | 3.3 [2.6 to 4.1] | 3.3 [2.6 to 4.3] | 2.8 [2.2 to 3.6] | 3.1 [2.5 to 3.9]

8. Secondary Outcome: Number of Seroprotected Subjects Against 3 Strains of Influenza Disease
Description: A seroprotected subject was defined as a vaccinated subject with serum Hemagglutination Inhibition (HI) titer ≥ 1:40. The 3 flu strains assessed were A/New Caledonia (H1N1), A/New York (H3N2) and B/Jiangsu (B).
Time Frame: At Day 0 and at Day 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 18-40 Y Group | Fluarix ≥65 Y Group | Fluarix-AS25 Group | Fluarix-AS50 Group | Fluarix- AS01B Group | Fluarix- AS01E Group
Number analyzed (Participants) | 75 | 49 | 74 | 75 | 75 | 75
Participants
  A/New Caledonia, Day 0 | 27 | 18 | 32 | 33 | 41 | 41
  A/New Caledonia, Day 21 | 75 | 35 | 67 | 74 | 73 | 70
  A/New York, Day 0 | 24 | 9 | 16 | 24 | 24 | 23
  A/New York, Day 21 | 70 | 40 | 70 | 70 | 72 | 70
  B/Jiangsu, Day 0 | 35 | 23 | 37 | 40 | 45 | 40
  B/Jiangsu, Day 21 | 75 | 46 | 71 | 74 | 75 | 73

9. Secondary Outcome: Number of Seroprotected Subjects Against 3 Strains of Influenza Disease
Description: as for outcome 8
Time Frame: At Day 90 and Day 180
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 18-40 Y Group | Fluarix ≥65 Y Group | Fluarix-AS25 Group | Fluarix-AS50 Group | Fluarix- AS01B Group | Fluarix- AS01E Group
Number analyzed (Participants) | 75 | 49 | 74 | 74 | 74 | 74
Participants
  A/New Caledonia, Day 90 | 75 | 37 | 66 | 68 | 71 | 69
  A/New Caledonia, Day 180: number analyzed (Participants) | 74 | 49 | 74 | 74 | 74 | 73
  A/New Caledonia, Day 180 | 72 | 34 | 58 | 62 | 60 | 62
  A/New York, Day 90 | 68 | 35 | 64 | 67 | 62 | 65
  A/New York, Day 180: number analyzed (Participants) | 74 | 49 | 74 | 74 | 74 | 73
  A/New York, Day 180 | 64 | 28 | 54 | 58 | 54 | 54
  B/Jiangsu, Day 90 | 71 | 47 | 66 | 72 | 72 | 67
  B/Jiangsu, Day 180: number analyzed (Participants) | 74 | 49 | 74 | 74 | 74 | 73
  B/Jiangsu, Day 180 | 67 | 41 | 63 | 70 | 69 | 63

10. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms.
Description: Assessed solicited local symptoms were haematoma, pain, redness and swelling. Any = occurrence of any local symptom regardless of intensity grade. Grade 3 pain = pain which prevented normal everyday activity. Grade 3 haematoma/redness/swelling = haematoma/redness/swelling spreading beyond 50 millimeters (mm).
Time Frame: During the 7-day (Days 0-6) follow-up period after vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects who received the vaccine dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 18-40 Y Group | Fluarix ≥65 Y Group | Fluarix-AS25 Group | Fluarix-AS50 Group | Fluarix- AS01B Group | Fluarix- AS01E Group
Number analyzed (Participants) | 75 | 50 | 75 | 75 | 75 | 75
Participants
  Haematoma, Any | 3 | 2 | 4 | 4 | 6 | 1
  Haematoma, > 50 mm | 0 | 0 | 1 | 0 | 0 | 0
  Pain, Any | 58 | 8 | 53 | 54 | 51 | 42
  Pain, Grade 3 | 0 | 0 | 1 | 1 | 2 | 0
  Redness, Any | 12 | 5 | 11 | 22 | 17 | 11
  Redness, > 50 mm | 0 | 0 | 3 | 9 | 5 | 4
  Swelling, Any | 9 | 1 | 14 | 15 | 12 | 9
  Swelling, > 50 mm | 0 | 0 | 5 | 6 | 4 | 3

11. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms.
Description: Assessed solicited general symptoms were fatigue, fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)], headache, joint pain, muscle aches and shivering. Any = occurrence of any general symptom regardless of intensity grade and relationship to vaccination. Grade 3 = symptoms that prevented normal activity. Grade 3 fever = fever >39°C. Related = general symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: During the 7-day (Days 0-6) follow-up period after vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects who received the vaccine dose.
Measure: Count of Participants; unit: Participants
Groups:
- Fluarix-AS01B Group: Subjects (aged ≥ 65 years) received 1 dose of the Fluarix vaccine adjuvanted with AS01B, administered intramuscularly in the deltoid region of the non-dominant arm.
- Fluarix-AS01E Group: Subjects (aged ≥ 65 years) received 1 dose of the Fluarix vaccine adjuvanted with AS01E, administered intramuscularly in the deltoid region of the non-dominant arm.
Arm/Group | Fluarix 18-40 Y Group | Fluarix ≥65 Y Group | Fluarix-AS25 Group | Fluarix-AS50 Group | Fluarix-AS01B Group | Fluarix-AS01E Group
Number analyzed (Participants) | 75 | 50 | 75 | 75 | 75 | 75
Participants
  Fatigue, Any | 34 | 7 | 31 | 34 | 31 | 22
  Fatigue, Grade 3 | 1 | 0 | 2 | 1 | 5 | 1
  Fatigue, Related | 26 | 7 | 27 | 34 | 31 | 19
  Fever (axillary), Any | 2 | 0 | 4 | 6 | 7 | 4
  Fever (axillary), Grade 3 | 0 | 0 | 1 | 1 | 0 | 0
  Fever (axillary), Related | 2 | 0 | 4 | 5 | 7 | 4
  Headache, Any | 24 | 12 | 28 | 27 | 21 | 14
  Headache, Grade 3 | 0 | 0 | 1 | 1 | 1 | 0
  Headache, Related | 17 | 8 | 26 | 25 | 20 | 14
  Joint pain, Any | 5 | 4 | 19 | 13 | 23 | 17
  Joint pain, Grade 3 | 0 | 0 | 1 | 0 | 1 | 1
  Joint pain, Related | 4 | 2 | 17 | 12 | 20 | 14
  Muscle aches, Any | 14 | 3 | 25 | 25 | 26 | 21
  Muscle aches, Grade 3 | 0 | 0 | 1 | 1 | 3 | 2
  Muscle aches, Related | 11 | 2 | 24 | 25 | 25 | 18
  Shivering, Any | 6 | 3 | 18 | 21 | 27 | 13
  Shivering, Grade 3 | 0 | 0 | 1 | 2 | 3 | 2
  Shivering, Related | 4 | 2 | 18 | 20 | 27 | 13

12. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs).
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 =event that prevented normal everyday activity. Related = event assessed by the investigator as causally related to the study vaccination.
Time Frame: During the 21-day (Days 0-20) follow-up period after vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects who received the vaccine dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 18-40 Y Group | Fluarix ≥65 Y Group | Fluarix-AS25 Group | Fluarix-AS50 Group | Fluarix- AS01B Group | Fluarix- AS01E Group
Number analyzed (Participants) | 75 | 50 | 75 | 75 | 75 | 75
Participants
  Any AEs | 37 | 6 | 27 | 26 | 31 | 24
  Grade 3 AEs | 1 | 0 | 4 | 6 | 4 | 3
  Related AEs | 11 | 2 | 9 | 14 | 18 | 5

13. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs).
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (Day 0 - Day 180)
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects who received the vaccine dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 18-40 Y Group | Fluarix ≥65 Y Group | Fluarix-AS25 Group | Fluarix-AS50 Group | Fluarix-AS01B Group | Fluarix-AS01E Group
Number analyzed (Participants) | 75 | 50 | 75 | 75 | 75 | 75
Participants | 0 | 3 | 5 | 6 | 4 | 6

ADVERSE EVENTS:
Time Frame: Unsolicited AEs: during the 21-day (Days 0-20) post-vaccination period; SAEs: during the entire study period (Days 0-180).
Description: For the solicited local and general symptoms occurring during the 7-day (Days 0-6) post-vaccination period, please refer to outcome measures 10 and 11 from the Outcome Measures section above.
Arm/Group | Fluarix 18-40 Y Group | Fluarix ≥65 Y Group | Fluarix-AS25 Group | Fluarix-AS50 Group | Fluarix- AS01B Group | Fluarix- AS01E Group
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/50 | 0/75 | 0/75 | 0/75 | 1/75
Serious Adverse Events (participants affected / at risk) | 0/75 | 3/50 | 5/75 | 6/75 | 4/75 | 6/75
Other Adverse Events (participants affected / at risk) | 37/75 | 6/50 | 27/75 | 26/75 | 31/75 | 24/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluarix 18-40 Y Group (N=75) | Fluarix ≥65 Y Group (N=50) | Fluarix-AS25 Group (N=75) | Fluarix-AS50 Group (N=75) | Fluarix- AS01B Group (N=75) | Fluarix- AS01E Group (N=75)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 2
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Transient ischemic attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluarix 18-40 Y Group (N=75) | Fluarix ≥65 Y Group (N=50) | Fluarix-AS25 Group (N=75) | Fluarix-AS50 Group (N=75) | Fluarix- AS01B Group (N=75) | Fluarix- AS01E Group (N=75)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 4
Influenza-like illness (General disorders) | 3 | 1 | 1 | 0 | 4 | 2
Nasopharyngitis (Infections and infestations) | 5 | 1 | 3 | 2 | 3 | 2
Headache (Nervous system disorders) | 10 | 0 | 1 | 0 | 1 | 3
Dysmenorrhoea (Reproductive system and breast disorders) | 4 | 0 | 0 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 2 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 1 | 2 | 2 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Injection site discolouration (General disorders) | 0 | 0 | 1 | 0 | 1 | 0
Injection site induration (General disorders) | 0 | 0 | 1 | 0 | 1 | 0
Injection site irritation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Injection site pruritus (General disorders) | 1 | 1 | 0 | 0 | 1 | 0
Injection site reaction (General disorders) | 2 | 1 | 1 | 0 | 2 | 0
Injection site warmth (General disorders) | 0 | 0 | 0 | 1 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0 | 2 | 1 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 3 | 0
Campylobacter infeection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1
Rhinitis (Infections and infestations) | 2 | 2 | 2 | 1 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 2 | 3 | 1 | 1
Urinary tract infections (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 2 | 0
Listless (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Scrotal ulcer (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 1 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.